CLINICAL TRIAL: NCT06662656
Title: ED50 of Sufentanil with Dexmedetomidine Analgesia During Laparoscopic Cholecystectomy
Brief Title: ED50 of Sufentanil for Intraoperative Analgesia
Acronym: ED50
Status: Not yet recruiting | Type: Observational
Sponsor: China International Neuroscience Institution (Other)
Responsible Party: Sponsor
Other Study IDs: CINI-AD-202403-13; CINI-AD-202403-13 (Other: XuanWu Hospital)
Record Dates: First submitted 2024-03-17; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Laparoscopic Cholecystectomy; Analgesics，Opioid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- 1μg/ kg group: Administration method of sufentanil: the dose of the first patient is 1μg / kg, and the ratio between adjacent doses is 1.2. ( IOC2 values of < 60, which were the target of this study, indicate adequate analgesic efect and analgesic level for regional surgery. IOC2 values of ≥ 60 indicate inadequate use of analgesics. If the analgesic effect of this patient is satisfactory, the next patient will use the lower dose. If the analgesic efect of this patient is not satisfactory, the next patient will use a higher dose. Starting from the first case of dissatisfaction, the number of observation units is counted. Dissatisfaction - satisfaction occurs at 7 exchange points and then the test ends.)
- 0.83μg/ kg group: Administration method of sufentanil: the dose of the first patient is 1μg / kg, and the ratio between adjacent doses is 1.2. 1/1.2=0.833 ( IOC2 values of < 60, which were the target of this study, indicate adequate analgesic efect and analgesic level for regional surgery. IOC2 values of ≥ 60 indicate inadequate use of analgesics. If the analgesic effect of this patient is satisfactory, the next patient will use the lower dose. If the analgesic efect of this patient is not satisfactory, the next patient will use a higher dose. Starting from the first case of dissatisfaction, the number of observation units is counted. Dissatisfaction - satisfaction occurs at 7 exchange points and then the test ends.)
- 0.69μg/ kg group: Administration method of sufentanil: the dose of the first patient is 1μg / kg, and the ratio between adjacent doses is 1.2. 0.833/1.2=0.694( IOC2 values of < 60, which were the target of this study, indicate adequate analgesic efect and analgesic level for regional surgery. IOC2 values of ≥ 60 indicate inadequate use of analgesics. If the analgesic effect of this patient is satisfactory, the next patient will use the lower dose. If the analgesic efect of this patient is not satisfactory, the next patient will use a higher dose. Starting from the first case of dissatisfaction, the number of observation units is counted. Dissatisfaction - satisfaction occurs at 7 exchange points and then the test ends.)
- 0.58μg/ kg group: Administration method of sufentanil: the dose of the first patient is 1μg / kg, and the ratio between adjacent doses is 1.2. 0.694/1.2=0.578( IOC2 values of < 60, which were the target of this study, indicate adequate analgesic efect and analgesic level for regional surgery. IOC2 values of ≥ 60 indicate inadequate use of analgesics. If the analgesic effect of this patient is satisfactory, the next patient will use the lower dose. If the analgesic efect of this patient is not satisfactory, the next patient will use a higher dose. Starting from the first case of dissatisfaction, the number of observation units is counted. Dissatisfaction - satisfaction occurs at 7 exchange points and then the test ends.)
- 0.48μg/ kg group: Administration method of sufentanil: the dose of the first patient is 1μg / kg, and the ratio between adjacent doses is 1.2. 0.578/1.2=0.482( IOC2 values of < 60, which were the target of this study, indicate adequate analgesic efect and analgesic level for regional surgery. IOC2 values of ≥ 60 indicate inadequate use of analgesics. If the analgesic effect of this patient is satisfactory, the next patient will use the lower dose. If the analgesic efect of this patient is not satisfactory, the next patient will use a higher dose. Starting from the first case of dissatisfaction, the number of observation units is counted. Dissatisfaction - satisfaction occurs at 7 exchange points and then the test ends.)
- 0.4μg/ kg group: Administration method of sufentanil: the dose of the first patient is 1μg / kg, and the ratio between adjacent doses is 1.2. 0.482/1.2=0.402( IOC2 values of < 60, which were the target of this study, indicate adequate analgesic efect and analgesic level for regional surgery. IOC2 values of ≥ 60 indicate inadequate use of analgesics. If the analgesic effect of this patient is satisfactory, the next patient will use the lower dose. If the analgesic efect of this patient is not satisfactory, the next patient will use a higher dose. Starting from the first case of dissatisfaction, the number of observation units is counted. Dissatisfaction - satisfaction occurs at 7 exchange points and then the test ends.)

SUMMARY:
1. Sufentanil as an strong analgesic is used widespreadly during laparoscopic cholecystectomy.
2. Lower dosages of sufentanil facilitated with dexmedetomidine can offer enough analgesia effect.
3. The investigator are planning use the most classical method for determining the ED50 or half effective concentration of sufentanil facilitated with dexmedetomidine using sequential method, which is also called" up and down method" and" ladder method".

DETAILED DESCRIPTION:
The concordance of the current research is that lower dosages of sufentanil facilitated with dexmedetomidine can offer enough analgesia effect through operation. However, the dosages of sufentanil used in various researches vary greatly of operations. Previous studies have shown that the amount of sufentanil required for intraoperative analgesia is smaller than that required while dexmedetomindine facilitated. Although the appropriate dosage of sufentanil required for operation can ensure the analgesic effect of operation, excessive dosage can cause severe choking during intubation, postoperative nausea and vomiting, hyperalgesia, and chronic postoperative pain. The investigator planning use the most classical method for determining the ED50 or half effective concentration of sufentainl combined with dexmedetomidine using sequential method, which is also called " up and down method" and " ladder method".

ELIGIBILITY:
Inclusion Criteria:

1. ASA I ~ II level;
2. BMI22-30kg/m2;
3. Those who intend to undergo laparoscopic cholecystectomy;
4. Age 18~65 years.

Exclusion Criteria:

1. Has been allergic to the drugs used in this study;
2. Patients with a history of chronic use of alcohol, smoke or other sedative drugs;
3. Patients took opioids and other analgesics before surgery;
4. Emergency operation;
5. Stress, anxiety resulting in secretion of catecholamine;
6. Patients with neuropsychiatric disorders, coma, depression, cognitive impairment and Alzheimer's disease;
7. Patients with epilepsy, autonomic nervous dysfunction and other diseases with abnormal EEG results;
8. SBP< 85 mmHg or HR< 45次/min;
9. Has implanted pacemaker;
10. Patients were unwilling or disable to finish whole study;
11. Patients with acute upper respiratory infections, liver or kidney failure and severe cardiopulmonary dysfunction.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in Xuanwu Hospital for elective laparoscopic cholecystectomy are selected. Before surgery, visitors recorded basic information such as the patient's sex, age, BMI, ASA grade in the ward.
Sampling Method: Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
The rate of the IOC2 target a reachment | through study completion, an average of 1 day
  The primary endpoint of the study was the attainment rate of the IOC2 target during operation

SECONDARY OUTCOMES:
visual analog scale score | 12 hours and 24hours after surgery
  visual analog scale (VAS) score at 12 h and 24 hours after operation,
The ratio of vomiting | 0 day, 1 day, 2 day after operation
  the ratio of vomiting
Systolic Blood Pressure | 0 day
  Systolic Blood Pressure reflect haemodynamics changeduring operation
Dystolic Blood Pressure | 0 day
  Dystolic Blood Pressure during operation
Mean Blood Pressure | 0 day
  Mean Blood Pressure during opeation
Heart rate | 0 day
  Heart rate during operation

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu hospital, Beijing, Beijing Municipality, China